CLINICAL TRIAL: NCT02301624
Title: A Phase III, Open-label Extension Trial of ECU-MG-301 to Evaluate the Safety and Efficacy of Eculizumab in Subjects With Refractory Generalized Myasthenia Gravis (gMG)
Brief Title: Extension Study of ECU-MG-301 to Evaluate Safety and Efficacy of Eculizumab in Refractory Generalized Myasthenia Gravis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECU-MG-302; 2013-002191-41 (EudraCT Number)
Record Dates: First submitted 2014-11-22; First posted 2014-11-26 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Refractory Generalized Myasthenia Gravis
Keywords: gMG; Myasthenia Gravis; safety; efficacy
MeSH Terms: conditions — Myasthenia Gravis | interventions — eculizumab

STUDY DESIGN:
Intervention Model Description: Following the Blind Induction Phase, all participants received open-label eculizumab.
Masking Description: The study consisted of a 4-week Blind Induction Phase to preserve the blinded nature of Study ECU-MG-301, followed by an Open-Label Maintenance Phase.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eculizumab/Eculizumab (Experimental): Blind Induction Phase: Participants who had received blinded treatment with eculizumab in Study ECU-MG-301 were administered eculizumab (4 vials/1200 milligrams [mg]) on Day 1 and Week 2 and placebo (4 vials/0 mg) at Weeks 1 and 3.
  Open-Label Maintenance Phase: Participants received open-label eculizumab (4 vials/1200 mg) every 2 weeks starting at Week 4 and continued throughout the study.
  Eculizumab 1200 mg was administered for up to 4 years in this extension study.
  Interventions: Biological: Eculizumab; Drug: Placebo
- Placebo/Eculizumab (Experimental): Blind Induction Phase: Participants who had received blinded treatment with placebo in Study ECU-MG-301 were administered eculizumab/placebo (3 vials/900 mg, plus 1 vial/0 mg, respectively) on Day 1 and Weeks 1 through 3.
  Open-Label Maintenance Phase: Participants received open-label eculizumab (4 vials/1200 mg) every 2 weeks starting at Week 4 and continued throughout the study.
  Eculizumab 1200 mg was administered for up to 4 years in this extension study.
  Interventions: Biological: Eculizumab; Drug: Placebo

INTERVENTIONS:
Biological: Eculizumab — Intravenous administration of eculizumab.
Drug: Placebo — Intravenous administration of matching placebo. Participants received placebo only during the Blind Induction Phase.

SUMMARY:
To evaluate the safety and efficacy of eculizumab in the treatment of refractory generalized myasthenia gravis (gMG) as an extension study for the participants who previously completed Study ECU-MG-301(NCT01997229).

DETAILED DESCRIPTION:
ECU-MG-302 was an extension study designed to provide the participants who completed Study ECU-MG-301 an opportunity to receive eculizumab and collect clinical data to provide long-term safety and efficacy information on eculizumab in participants with refractory gMG.

After receiving blinded study treatment (eculizumab or placebo) in Study ECU-MG-301 for 26 weeks, participants were eligible to enroll in the ECU-MG-302 extension study. Participants were to enter Study ECU-MG-302 within 2 weeks after completing their Week 26 visit in Study ECU-MG-301.

Study ECU-MG-302 consisted of a 4-week Blind Induction Phase to preserve the blinded nature of Study ECU-MG-301, an Open-Label Maintenance Phase (up to 4 years), and a Safety Follow-up visit 8 weeks after the last dose for participants who withdrew from the study or discontinued eculizumab treatment at any time and for any reason after receiving any amount of eculizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has completed Study ECU-MG-301.
2. Participant has given written informed consent.
3. Participant was willing and able to comply with the protocol requirements for the duration of the study.
4. Female participant of childbearing potential must have had a negative pregnancy test (serum human chorionic gonadotropin). All participants were required to practice an effective, reliable, and medically approved contraceptive regimen during the study and for up to 5 months following discontinuation of treatment.

Exclusion Criteria:

1. Participants who withdrew from Study ECU-MG-301 as a result of an adverse event related to study drug.
2. Female participants who were pregnant, breastfeeding, or intended to conceive during the course of the study.
3. Unresolved meningococcal infection
4. Hypersensitivity to murine proteins or to one of the excipients of eculizumab
5. Any medical condition or circumstances that, in the opinion of the investigator, might have interfered with the participant's participation in the study, posed any added risk for the participant, or confounded the assessment of the participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2014-11-12 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Yountz, MD, Study Director — Alexion Pharmaceuticals, Inc.
Locations (59):
- United States (25):
  - Birmingham, Alabama
  - Los Angeles, California
  - Orange, California
  - Palo Alto, California
  - San Francisco, California
  - New Haven, Connecticut
  - Jacksonville, Florida
  - Miami, Florida
  - Tampa, Florida
  - Springfield, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - Las Vegas, Nevada
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Columbus, Ohio
  - Portland, Oregon
  - San Antonio, Texas
  - Burlington, Vermont
  - Seattle, Washington
- Buenos Aires, Argentina
- Belgium (3):
  - Edegem
  - Ghent
  - Leuven
- São Paulo, Brazil
- Edmonton, Canada
- Czechia (2):
  - Ostrava - Poruba
  - Prague
- Denmark (2):
  - Arhus C
  - Copenhagen
- Turku, Finland
- Szeged, Hungary
- Italy (3):
  - Milan
  - Napoli
  - Roma
- Japan (8):
  - Chiba
  - Fukuoka
  - Hanamaki
  - Hokkaido
  - Miyagi
  - Nagasaki
  - Osaka
  - Osaka-Fu
- Amsterdam, Netherlands
- Seoul, South Korea
- Spain (2):
  - Barcelona
  - Madrid
- Stockholm, Sweden
- Turkey (Türkiye) (3):
  - Ankara
  - Izmir
  - Kocaeli
- United Kingdom (3):
  - Birmingham
  - Liverpool
  - London

REFERENCES:
- [Result] Muppidi S, Utsugisawa K, Benatar M, Murai H, Barohn RJ, Illa I, Jacob S, Vissing J, Burns TM, Kissel JT, Nowak RJ, Andersen H, Casasnovas C, de Bleecker JL, Vu TH, Mantegazza R, O'Brien FL, Wang JJ, Fujita KP, Howard JF Jr; Regain Study Group. Long-term safety and efficacy of eculizumab in generalized myasthenia gravis. Muscle Nerve. 2019 Jul;60(1):14-24. doi: 10.1002/mus.26447. Epub 2019 Mar 8. PMID 30767274
- [Result] Andersen H, Mantegazza R, Wang JJ, O'Brien F, Patra K, Howard JF Jr; REGAIN Study Group. Correction to: Eculizumab improves fatigue in refractory generalized myasthenia gravis. Qual Life Res. 2019 Aug;28(8):2255. doi: 10.1007/s11136-019-02204-x. PMID 31115842
- [Result] Andersen H, Mantegazza R, Wang JJ, O'Brien F, Patra K, Howard JF Jr; REGAIN Study Group. Eculizumab improves fatigue in refractory generalized myasthenia gravis. Qual Life Res. 2019 Aug;28(8):2247-2254. doi: 10.1007/s11136-019-02148-2. Epub 2019 Mar 23. PMID 30905021
- [Result] Murai H, Uzawa A, Suzuki Y, Imai T, Shiraishi H, Suzuki H, Okumura M, O'Brien F, Wang JJ, Fujita KP, Utsugisawa K; REGAIN Study Group. Long-term efficacy and safety of eculizumab in Japanese patients with generalized myasthenia gravis: A subgroup analysis of the REGAIN open-label extension study. J Neurol Sci. 2019 Dec 15;407:116419. doi: 10.1016/j.jns.2019.08.004. Epub 2019 Aug 3. PMID 31698177
- [Derived] Siddiqi ZA, Nowak RJ, Mozaffar T, O'Brien F, Yountz M, Patti F; REGAIN Study Group. Eculizumab in refractory generalized myasthenia gravis previously treated with rituximab: subgroup analysis of REGAIN and its extension study. Muscle Nerve. 2021 Dec;64(6):662-669. doi: 10.1002/mus.27422. Epub 2021 Oct 14. PMID 34590717
- [Derived] Murai H, Suzuki S, Hasebe M, Fukamizu Y, Rodrigues E, Utsugisawa K. Safety and effectiveness of eculizumab in Japanese patients with generalized myasthenia gravis: interim analysis of post-marketing surveillance. Ther Adv Neurol Disord. 2021 Mar 16;14:17562864211001995. doi: 10.1177/17562864211001995. eCollection 2021. PMID 33796147
- [Derived] Nowak RJ, Muppidi S, Beydoun SR, O'Brien FL, Yountz M, Howard JF Jr. Concomitant Immunosuppressive Therapy Use in Eculizumab-Treated Adults With Generalized Myasthenia Gravis During the REGAIN Open-Label Extension Study. Front Neurol. 2020 Nov 24;11:556104. doi: 10.3389/fneur.2020.556104. eCollection 2020. PMID 33329303
- [Derived] Mantegazza R, Wolfe GI, Muppidi S, Wiendl H, Fujita KP, O'Brien FL, Booth HDE, Howard JF Jr; REGAIN Study Group. Post-intervention Status in Patients With Refractory Myasthenia Gravis Treated With Eculizumab During REGAIN and Its Open-Label Extension. Neurology. 2021 Jan 26;96(4):e610-e618. doi: 10.1212/WNL.0000000000011207. Epub 2020 Nov 23. PMID 33229455
- [Derived] Mantegazza R, O'Brien FL, Yountz M, Howard JF Jr; REGAIN study group. Consistent improvement with eculizumab across muscle groups in myasthenia gravis. Ann Clin Transl Neurol. 2020 Aug;7(8):1327-1339. doi: 10.1002/acn3.51121. Epub 2020 Jul 22. PMID 32700461
- [Derived] Jacob S, Murai H, Utsugisawa K, Nowak RJ, Wiendl H, Fujita KP, O'Brien F, Howard JF Jr. Response to eculizumab in patients with myasthenia gravis recently treated with chronic IVIg: a subgroup analysis of REGAIN and its open-label extension study. Ther Adv Neurol Disord. 2020 May 6;13:1756286420911784. doi: 10.1177/1756286420911784. eCollection 2020. PMID 32426038
- [Derived] Vissing J, Jacob S, Fujita KP, O'Brien F, Howard JF; REGAIN study group. 'Minimal symptom expression' in patients with acetylcholine receptor antibody-positive refractory generalized myasthenia gravis treated with eculizumab. J Neurol. 2020 Jul;267(7):1991-2001. doi: 10.1007/s00415-020-09770-y. Epub 2020 Mar 18. PMID 32189108

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed Study ECU-MG-301 (NCT01997229) were eligible to participate in Study ECU-MG-302.
Period: Blind Induction Phase
Arm/Group | Eculizumab/Eculizumab | Placebo/Eculizumab
Started | 56 | 61
Received at Least 1 Dose of Study Drug | 56 | 61
Completed | 55 | 61
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Open-label Maintenance Phase
Arm/Group | Eculizumab/Eculizumab | Placebo/Eculizumab
Started | 55 | 61
Received at Least 1 Dose of Study Drug | 55 | 61
Completed | 43 | 44
Not Completed | 12 | 17
Not completed — Withdrawal by Subject | 4 | 8
Not completed — Adverse Event | 2 | 5
Not completed — Physician Decision | 3 | 3
Not completed — Death | 2 | 1
Not completed — Participant felt no change in condition | 1 | 0

BASELINE CHARACTERISTICS:
Population: All eligible enrolled participants who received at least 1 dose of study drug in this extension study.
Groups:
- Eculizumab/Eculizumab: Blind Induction Phase: Participants who had received blinded treatment with eculizumab in Study ECU-MG-301 were administered eculizumab (4 vials/1200 mg) on Day 1 and Week 2 and placebo (4 vials/0 mg) at Weeks 1 and 3.
  Open-Label Maintenance Phase: Participants received open-label eculizumab (4 vials/1200 mg) every 2 weeks starting at Week 4 and continued throughout the study.
  Eculizumab 1200 mg was administered for up to 4 years in this extension study.
- Total: Total of all reporting groups
Arm/Group | Eculizumab/Eculizumab | Placebo/Eculizumab | Total
Number analyzed (Participants) | 56 | 61 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (15.52) | 47.5 (17.85) | 47.4 (16.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 41 | 79
  Male | 18 | 20 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 18
  Not Hispanic or Latino | 45 | 48 | 93
  Unknown or Not Reported | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 16 | 19
  Black or African American | 0 | 2 | 2
  White | 47 | 41 | 88
  Multiple | 1 | 0 | 1
  Unknown | 1 | 0 | 1
  Other | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Count Of Participants With Treatment-Emergent Adverse Events
Description: Treatment-emergent adverse events (TEAEs) are adverse events with onset on or after the first study drug dose in Study ECU-MG-302. Likewise, treatment-emergent serious adverse events (TESAEs) are serious adverse events that onset on or after the first study drug dose in Study ECU-MG-302. A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Day 1 (after dosing) through End of Study (Week 208)
Population: All participants who received at least 1 dose of eculizumab in this extension study.
Measure: Count of Participants; unit: Participants
Groups:
- Eculizumab/Eculizumab: After receiving blinded treatment with eculizumab in Study ECU-MG-301 for 26 weeks, all participants received blinded study drug weekly for 4 weeks, then received open-label eculizumab 1200 mg every 2 weeks for up to 4 years in this extension study.
- Placebo/Eculizumab: After receiving blinded treatment with placebo in Study ECU-MG-301 for 26 weeks, all participants received blinded study drug weekly for 4 weeks, then received open-label eculizumab 1200 mg every 2 weeks for up to 4 years in this extension study.
Arm/Group | Eculizumab/Eculizumab | Placebo/Eculizumab
Number analyzed (Participants) | 56 | 61
Participants
  TEAEs | 55 | 59
  TEAEs leading to withdrawal | 3 | 5
  TESAEs | 30 | 30
  TESAEs leading to withdrawal | 3 | 4
  Deaths | 2 | 1

2. Secondary Outcome: Change From Baseline In Myasthenia Gravis Activities Of Daily Living Profile (MG-ADL) Total Score At Week 4 And Week 130
Description: The MG-ADL scale is a validated 8-item patient-reported outcome measure. Participants assessed their functional disability secondary to ocular (2 items), bulbar (3 items), respiratory (1 item), and gross motor or limb impairment (2 items). These 8 items were not weighted and were individually graded from 0 (normal) to 3 (most severe), providing a total MG-ADL score ranging from 0 to 24 points. A reduction in score indicates improvement in condition. Baseline was defined as the last available assessment prior to treatment (first study drug infusion) with eculizumab in Study ECU-MG-302. Change from Baseline in MG-ADL total score at Week 4 (blind induction phase) and at Week 130 (open-label eculizumab phase) are presented.
Time Frame: Baseline, Week 4 and Week 130
Population: All participants who received at least 1 dose of eculizumab in this extension study and had an MG-ADL efficacy assessment after study drug infusion at the specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eculizumab/Eculizumab | Placebo/Eculizumab
Number analyzed (Participants) | 55 | 61
units on a scale
  Change from Baseline At Week 4 (Blind Induction) | -0.2 (1.77) | -2.4 (3.04)
  Change from Baseline at Week 130 (Open-label): number analyzed (Participants) | 35 | 36
  Change from Baseline at Week 130 (Open-label) | -0.7 (4.19) | -3.9 (3.68)

ADVERSE EVENTS:
Time Frame: Day 1 after dosing of study drug through Week 208.
Description: All eligible enrolled participants who received at least 1 dose of study drug.
Groups:
- Eculizumab (Combined Total): All participants who received at least 1 dose of eculizumab in the extension study. Participants received open-label eculizumab (4 vials/1200 mg) every 2 weeks starting at Week 4 and continued throughout the study.
  Eculizumab 1200 mg was administered for up to 4 years in this extension study.
Arm/Group | Eculizumab/Eculizumab | Placebo/Eculizumab | Eculizumab (Combined Total)
All-Cause Mortality (participants affected / at risk) | 2/56 | 1/61 | 3/117
Serious Adverse Events (participants affected / at risk) | 30/56 | 30/61 | 60/117
Other Adverse Events (participants affected / at risk) | 54/56 | 59/61 | 113/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Eculizumab/Eculizumab (N=56) | Placebo/Eculizumab (N=61) | Eculizumab (Combined Total) (N=117)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 1
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 1
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 1
Chest pain (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 3 | 0 | 3
Chronic hepatic failure (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 1
Autoimmune disorder (Immune system disorders) | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 1
Aspergillus infection (Infections and infestations) | 1 | 0 | 1
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 2
Bursitis infective staphylococcal (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 1
Colonic abscess (Infections and infestations) | 1 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 1
Device related sepsis (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 2 | 3
Influenza (Infections and infestations) | 2 | 0 | 2
Localised infection (Infections and infestations) | 1 | 1 | 2
Meningitis meningococcal (Infections and infestations) | 1 | 0 | 1
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 2 | 4
Pseudomonal sepsis (Infections and infestations) | 1 | 0 | 1
Pseudomonas infection (Infections and infestations) | 1 | 0 | 1
Rectal abscess (Infections and infestations) | 1 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 1
Sepsis (Infections and infestations) | 2 | 1 | 3
Tonsillitis (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 2 | 2
Wound infection (Infections and infestations) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 1 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 1 | 0 | 1
Central obesity (Metabolism and nutrition disorders) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/18 | 1/20 | 1/38 — Adverse event affects male participants only
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 2 | 3
Loss of consciousness (Nervous system disorders) | 0 | 1 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 1
Myasthenia gravis (Nervous system disorders) | 7 | 9 | 16
Myasthenia gravis crisis (Nervous system disorders) | 2 | 2 | 4
Quadriparesis (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0/38 | 1/41 | 1/79 — Adverse event affects female participants only
Ovarian cyst (Reproductive system and breast disorders) | 1/38 | 0/41 | 1/79 — Adverse event affects female participants only
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/38 | 0/41 | 1/79 — Adverse event affects female participants only
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Extremity necrosis (Vascular disorders) | 0 | 1 | 1
Haematoma (Vascular disorders) | 0 | 1 | 1
Lupus vasculitis (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Eculizumab/Eculizumab (N=56) | Placebo/Eculizumab (N=61) | Eculizumab (Combined Total) (N=117)
Anaemia (Blood and lymphatic system disorders) | 5 | 3 | 8
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 2 | 5
Lymphopenia (Blood and lymphatic system disorders) | 3 | 0 | 3
Atrial fibrillation (Cardiac disorders) | 4 | 1 | 5
Palpitations (Cardiac disorders) | 1 | 4 | 5
Tachycardia (Cardiac disorders) | 4 | 2 | 6
Ear pain (Ear and labyrinth disorders) | 2 | 4 | 6
Vertigo (Ear and labyrinth disorders) | 3 | 4 | 7
Cataract (Eye disorders) | 4 | 5 | 9
Dry eye (Eye disorders) | 2 | 4 | 6
Eye pain (Eye disorders) | 0 | 4 | 4
Abdominal discomfort (Gastrointestinal disorders) | 4 | 6 | 10
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 5
Abdominal pain upper (Gastrointestinal disorders) | 2 | 6 | 8
Dental caries (Gastrointestinal disorders) | 2 | 5 | 7
Diarrhoea (Gastrointestinal disorders) | 15 | 14 | 29
Dyspepsia (Gastrointestinal disorders) | 2 | 4 | 6
Nausea (Gastrointestinal disorders) | 9 | 13 | 22
Tooth disorder (Gastrointestinal disorders) | 3 | 0 | 3
Toothache (Gastrointestinal disorders) | 3 | 5 | 8
Vomiting (Gastrointestinal disorders) | 3 | 7 | 10
Chest pain (General disorders) | 4 | 2 | 6
Fatigue (General disorders) | 8 | 7 | 15
Influenza like illness (General disorders) | 4 | 3 | 7
Oedema peripheral (General disorders) | 4 | 3 | 7
Peripheral swelling (General disorders) | 3 | 2 | 5
Pyrexia (General disorders) | 5 | 8 | 13
Seasonal allergy (Immune system disorders) | 3 | 7 | 10
Bronchitis (Infections and infestations) | 6 | 7 | 13
Cellulitis (Infections and infestations) | 4 | 4 | 8
Gastroenteritis (Infections and infestations) | 6 | 5 | 11
Gastroenteritis viral (Infections and infestations) | 4 | 6 | 10
Herpes zoster (Infections and infestations) | 3 | 1 | 4
Influenza (Infections and infestations) | 11 | 10 | 21
Nasopharyngitis (Infections and infestations) | 20 | 22 | 42
Oral herpes (Infections and infestations) | 3 | 3 | 6
Pharyngitis (Infections and infestations) | 3 | 0 | 3
Pneumonia (Infections and infestations) | 4 | 6 | 10
Respiratory tract infection (Infections and infestations) | 4 | 0 | 4
Sinusitis (Infections and infestations) | 7 | 4 | 11
Tonsillitis (Infections and infestations) | 1 | 4 | 5
Upper respiratory tract infection (Infections and infestations) | 12 | 15 | 27
Urinary tract infection (Infections and infestations) | 10 | 8 | 18
Contusion (Injury, poisoning and procedural complications) | 7 | 5 | 12
Fall (Injury, poisoning and procedural complications) | 8 | 6 | 14
Infusion related reaction (Injury, poisoning and procedural complications) | 4 | 7 | 11
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 2 | 5
Procedural pain (Injury, poisoning and procedural complications) | 2 | 4 | 6
Rib fracture (Injury, poisoning and procedural complications) | 3 | 0 | 3
Tooth fracture (Injury, poisoning and procedural complications) | 3 | 1 | 4
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 4
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 | 2 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 12 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 7 | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 6 | 11
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 7 | 12
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 8 | 17
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4 | 6
Dizziness (Nervous system disorders) | 3 | 6 | 9
Headache (Nervous system disorders) | 20 | 24 | 44
Migraine (Nervous system disorders) | 4 | 3 | 7
Myasthenia gravis (Nervous system disorders) | 12 | 5 | 17
Anxiety (Psychiatric disorders) | 4 | 4 | 8
Depression (Psychiatric disorders) | 3 | 8 | 11
Insomnia (Psychiatric disorders) | 7 | 2 | 9
Dysuria (Renal and urinary disorders) | 3 | 1 | 4
Ovarian cyst (Reproductive system and breast disorders) | 3/38 | 0/41 | 3/79 — Adverse event affects female participants only
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 10 | 22
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 9 | 12
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2 | 5
Eczema (Skin and subcutaneous tissue disorders) | 3 | 3 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 4 | 8
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 6
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 1 | 4
Hypertension (Vascular disorders) | 6 | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications at least 60 days prior to public release. Within 30 days of receipt, Sponsor shall advise of any information which is Confidential Information (other than Study Data) or which may impair the availability of patent protection for Inventions. Sponsor can require removal of specifically identified Confidential Information (other than Study Data) and/or delay the communication an additional 60 days to enable Sponsor to seek patent protection for Inventions.

DOCUMENTS (2):
  • Study Protocol (2016-12-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT02301624/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT02301624/SAP_001.pdf